CLINICAL TRIAL: NCT00030589
Title: A Muliticenter, Dose-Reandomized Evaluation Of Targretin Capsules Plus PUVA In Patients With Stage IB - IIA Cutaneous T-Cell Lymphoma
Brief Title: Chemotherapy and Photodynamic Therapy in Treating Patients With Cutaneous T-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Millennix (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069179; MILL-61896; LIGAND-MILL-61896; NU-IRB-837-002
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2003-10

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Bexarotene; Methoxsalen; Ultraviolet Therapy

INTERVENTIONS:
Drug: bexarotene
Drug: methoxsalen
Procedure: UV light therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill cancer cells. Photosensitizing drugs, such as methoxsalen, are absorbed by cancer cells and, when exposed to light, become active and kill the cancer cells. Combining chemotherapy with photodynamic therapy may be an effective treatment for cutaneous T-cell lymphoma.

PURPOSE: Randomized phase II trial to study the effectiveness of combining different doses of bexarotene with photodynamic therapy in treating patients who have stage IB or stage IIA cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of 2 different doses of bexarotene administered with ultraviolet A light therapy with methoxsalen (PUVA) in patients with stage IB or IIA cutaneous T-cell lymphoma.
* Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive a lower dose of oral bexarotene once daily on weeks 1-26. Patients also receive ultraviolet A light therapy with oral methoxsalen 3 times weekly on weeks 2-26.
* Arm II: Patients receive a higher dose of oral bexarotene once daily on weeks 1-26. Patients also receive ultraviolet A light therapy as in arm I.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma within the past year
* Stage IB or IIA disease

  * No prior diagnosis more advanced than stage IIA disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 9 g/dL
* WBC at least 2,000/mm^3
* Absolute lymphocyte count normal

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* No significant hepatic dysfunction

Renal:

* Creatinine no greater than 2 times ULN
* Calcium no greater than 11.5 mg/dL
* No significant renal dysfunction

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 1 month after study participation
* Fasting triglycerides normal (fenofibrate or another anti-lipemic agent allowed except gemfibrozil)
* HIV negative
* No other concurrent known serious medical illness or infection that would preclude study participation
* No prior uncontrolled hyperlipidemia
* No pancreatitis or clinically significant risk factors for developing pancreatitis
* No known allergy or sensitivity to retinoid class drugs or fenofibrate or idiosyncratic reactions to psoralen compounds
* No history of light-sensitive disease states (e.g., lupus, porphyria, or albinism) or aphakia
* No prior or concurrent melanoma or invasive squamous cell carcinoma
* No pre-existing gallbladder disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior systemic anticancer interferon
* No prior systemic anticancer denileukin diftitox

Chemotherapy:

* At least 30 days since prior topical anticancer carmustine or mechlorethamine
* No prior systemic anticancer alkaloid chemotherapy
* No other concurrent systemic or topical anticancer chemotherapy (e.g., methotrexate or cyclophosphamide)

Endocrine therapy:

* At least 30 days since prior topical anticancer corticosteroids
* No concurrent systemic or topical anticancer corticosteroids

Radiotherapy:

* No concurrent localized radiotherapy to specific study lesions except at investigator's discretion

Surgery:

* Not specified

Other:

* No prior systemic anticancer therapy
* At least 30 days since prior topical anticancer therapy (e.g., ultraviolet B light or psoralen-ultraviolet-light therapy)
* At least 30 days since prior participation in another investigational drug study
* At least 30 days since prior vitamin A (at doses of more than 15,000 IU/day) or other retinoid class drugs
* No other concurrent systemic or topical anticancer drugs or therapies
* No other concurrent systemic retinoid class drugs, beta-carotene compounds, or vitamin A (at doses of more than 15,000 IU/day)
* No other concurrent investigational medication
* No concurrent gemfibrozil
* No concurrent statin class anti-lipemics combined with fibrate class anti-lipemics (e.g., atorvastatin with fenofibrate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Joan Guitart, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (19):
- United States (19):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern University Medical Center, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Slidell, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - StonyBrook Dermatology Associates, P.C., East Setauket, New York
  - St. Luke's-Roosevelt Hospital Center - Roosevelt Division, New York, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Knoxville Dermatology Group, P.C., Knoxville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Tyler, Texas

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956